CLINICAL TRIAL: NCT04336852
Title: Development of a Clinically-relevant Test for Assessment of Cerebral Vascular Function
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Administratively Closed-PI left institution
Sponsor: University of Illinois at Chicago (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2020-0318; 1F32HL144082-01A1 (NIH); 5F32HL144082-02 (NIH)
Record Dates: First submitted 2020-04-01; First posted 2020-04-07 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Cerebrovascular Disorders; Cerebrovascular Disease
Keywords: brain blood flow; brain vascular function
MeSH Terms: conditions — Cerebrovascular Disorders

STUDY DESIGN:
Intervention Model Description: Three groups of subjects (young, older, cigarette smokers) complete the same intervention, in an independent-group design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm 1 (Experimental)
  Interventions: Procedure: Flow mediated dilation (brachial and femoral arteries); Procedure: Cerebral vascular reactivity to carbon dioxide (CO2); Procedure: Cerebral vascular function test

INTERVENTIONS:
Procedure: Flow mediated dilation (brachial and femoral arteries) — Assessment of vascular function of the brachial and femoral arteries.
Procedure: Cerebral vascular reactivity to carbon dioxide (CO2) — Cerebral blood flow responses to increasing partial pressure of CO2
Procedure: Cerebral vascular function test — Cerebral blood flow responses to a reactive hyperemia stimulus

SUMMARY:
The goal of this study is to develop a test of cerebral vessel function by inducing a reactive hyperemia that will elicit a rapid and profound increase in cerebral vessel shear stress. The results of this project may lead to development of a test with prognostic/predictive utility for individual risk assessment of a future cerebrovascular event/disease. This information will be of vital importance to the medical community in regards to cerebrovascular health in aging individuals, and testing of interventions and therapies that may ameliorate these effects.

ELIGIBILITY:
Inclusion Criteria:

Young and Older Healthy Adults:

* Males and females willing and able to provide informed consent
* Aged between 18-35 years (Young) or 60-80 years (Older)
* Premenopausal women will be tested within 1-4 days after menses begins to control for hormone status
* Women taking oral contraceptives will be allowed to participate and they will be tested in the low hormone or placebo phase
* Postmenopausal women (at least 12 months since last menstrual cycle) who are not on hormone replacement therapy will be eligible
* Sedentary or recreationally active
* Non-tobacco/nicotine users (e.g., cigarettes, chewing tobacco, nicotine gum or patches)
* Laboratory measured systolic blood pressure <140 mmHg and diastolic blood pressure <90 mmHg
* Normal 12-lead ECG (reviewed by a physician)
* Normal clinical results from a medical exam reviewed by a board certified physician (e.g., Medical & Behavioral Health Questionnaire - see attached document)
* Body mass index (BMI) <40 kg/m2 unless athletic/muscular build; calculation = body weight (kg)/height (m2); this criteria is used to ensure subjects will fit inside the LBNP chamber
* Females only: documentation of a negative pregnancy test prior to the familiarization and experimental sessions

Young and Older Chronic Smokers of Tobacco Cigarettes:

The same criteria (a-c and e-i above) as Young and Older Healthy Adults, except:

- Chronic smokers of tobacco cigarettes only (i.e., at least 20 pack year use)

Exclusion Criteria:

Young and Older Healthy Adults:

* Age <18 years, or 40-60 years, or >80 years
* Body mass index (BMI) >40 kg/m2 unless athletic/muscular build; calculation = body weight (kg)/height (m2)
* Regular tobacco/nicotine users within the last 6 months (e.g., cigarettes, chewing tobacco, nicotine gum or patches)
* Not abstaining from the following 24 hours prior to the familiarization session and the experimental session: exercise, alcoholic substances, prescription or non-prescription medications (unless cleared by the medical screener), dietary supplements, herbal medications, caffeinated substances (including coffee, tea (iced or hot), caffeinated energy drinks or sodas).
* Not fasted for at least 3-4 hours prior to the experimental sessions.
* Positive pregnancy test
* Hormone replacement therapy (males and females)
* Females with an erratic/irregular menstrual cycle
* Females who are using a continually-releasing hormonal (e.g., NuvaRing™ or other hormone-releasing vaginal rings, Depo Provera shot, birth control implants such as Nexplanon) and who do not have a regular menstrual cycle
* Use of prescription drugs, non-prescription drugs or herbal medicines known to alter autonomic function unless cleared prior to the study
* Any metabolic disease, except individuals who are on cholesterol-lowering medications (older subjects only; young subjects on cholesterol-lowering medications will be excluded)
* Use of two or more anti-hypertensive medications (older subjects only; young subjects on anti-hypertensive medications will be excluded)
* Use of beta blockers
* Frequent use of bronchodilators
* Use of anti-coagulant therapy
* Current or past history of hyperthyroidism, or other thyroid hormone-related disease
* Signs of cardiovascular abnormalities (e.g., resting systolic blood pressure >140 mmHg or diastolic blood pressure >90 mmHg; abnormal 12-lead ECG)
* History of cerebrovascular abnormalities (e.g., prior stroke, transient ischemic attacks, epilepsy)
* Known history of atherosclerosis of the carotid arteries (i.e., plaque formation)
* Known history of peripheral artery disease (PAD)
* Concussion and or other loss of consciousness within the past 30 days.
* Autonomic dysfunction (e.g., Shy-Drager Syndrome, Bradbury-Eggleston syndrome, sinus arrhythmia, idiopathic orthostatic hypotension, fainting disorder)
* Respiratory illnesses (e.g., chronic asthma (including exercise-induced asthma), Chronic Obstructive Pulmonary Disease, Reactive Airway Disease)
* History of anaphylaxis
* History of pre-syncopal/syncopal episodes or orthostatic hypotension
* Donated blood within the last 60 days
* History or family history of abnormal blood clotting, clots in deep veins in the legs or pelvis, or blood clots to the lungs
* Known or suspected abdominal hernia
* History of alcohol or drug abuse which inhibits the subject's ability to complete this study
* Known depression, anxiety, or any other mental health issue which inhibits the subject's ability to complete this study

Young and Older Chronic Smokers of Tobacco Cigarettes

The same criteria (a-b and d-dd above) as Young and Older Healthy Adults, except:

- Less than 20 pack year use of tobacco cigarettes, or regular use of other tobacco/nicotine products within the last 6 months (e.g., electronic cigarettes, chewing tobacco, nicotine gum or patches).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2018-09-14 (Actual); Primary Completion 2023-05-12 (Actual); Study Completion 2023-05-12 (Actual)

PRIMARY OUTCOMES:
Cerebral vascular function | 3-months
  Assessment of internal carotid artery dilation and blood flow in response to a reactive hyperemic stimulus
Cerebral vascular reactivity to carbon dioxide (CO2) | 3-months
  Assessment of blood flow (or velocity) through the internal carotid artery and middle cerebral artery with a standardized CO2 stimulus (+5 mmHg)
Flow mediated dilation (brachial and femoral arteries) | 3-months
  Assessment of artery dilation and blood flow in response to a reactive hyperemic stimulus

CONTACTS AND LOCATIONS:
Overall Officials: Alexander J Rosenberg, PhD, Principal Investigator — University of Illinois at Chicago
Locations (2):
- United States (2):
  - University of Illinois at Chicago, Chicago, Illinois
  - University of North Texas Health Science Center, Fort Worth, Texas

IPD SHARING:
Plan to Share IPD: No